CLINICAL TRIAL: NCT03078907
Title: A Multi-center, Double-blind, Placebo-controlled Phase 4 Study in Patients With Pulmonary Arterial Hypertension to Assess the Effect of Selexipag on Daily Life Physical Activity and Patient's Self-reported Symptoms and Their Impacts
Brief Title: Effect of Selexipag on Daily Life Physical Activity of Patients With Pulmonary Arterial Hypertension.
Acronym: TRACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-065A404
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: daily life; physical activity; actigraphy; PAH-SYMPACT
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Motor Activity | interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selexipag (Experimental): Selexipag is up-titrated from Day 1 to Week 12 to the individualized highest tolerated dose (HTD), which can range from 200 mcg b.i.d. to 1600 mcg b.i.d., in 200 mcg steps starting with 200 mcg b.i.d. Then, the dose is increased in increments of 200 mcg b.i.d., usually at weekly intervals, depending on the dose tolerability. Up-titration is followed by a stable maintenance treatment period at the highest tolerated dose, from Week 13 to Week 24.
  Interventions: Drug: Selexipag
- Placebo (Placebo Comparator): Regimen and titration scheme similar to those in the selexipag group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selexipag — Film-coated tablets for oral use; one tablet (200 mcg) to eight tablets (1600 mcg) are administered depending on the individual tolerability.
  Other Names: ACT-293987; Uptravi
  Arms: Selexipag
Drug: Placebo — Matching film coated tablets
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of selexipag on the physical activity of patients with pulmonary arterial hypertension (PAH) in their daily life, by using a wearable wrist device (actigraph). The actigraph will collect data on daily life physical activity in the patient's real environment. In addition, the PAH symptoms and their impacts will be assessed by using an electronic patient reported outcome measure in the patient's real environment. Patients will be assigned randomly to either selexipag or placebo.

DETAILED DESCRIPTION:
This study is designed as exploratory with the purpose to generate hypotheses on new endpoints

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years old inclusive.
* Women of childbearing potential must have a negative serum pregnancy test at planned visits and use an acceptable method of birth control from screening up to 30 days after study treatment discontinuation.
* Symptomatic pulmonary arterial hypertension (PAH) belonging to one of the following subgroups only:

  * Idiopathic
  * Heritable
  * Drug or toxin induced
  * Associated with one of the following: connective tissue disease; HIV infection; corrected simple congenital heart disease.
* With the following hemodynamic characteristics assessed by right heart catheterization (RHC) prior to randomization:

  * Mean pulmonary artery pressure (mPAP) ≥ 25 mmHg
  * Pulmonary vascular resistance (PVR) ≥ 240 dyn•sec/cm5 (or 3 Wood Units)
  * Pulmonary artery wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) ≤ 15 mmHg.
* Treatment with an endothelin receptor antagonist (ERA) for at least 90 days and on a stable dose for 30 days prior to randomization.
* If an ERA is given in combination with a phosphodiesterase-5 (PDE-5) inhibitor or soluble guanylate cyclase (sGC) stimulator, these treatments must be ongoing for at least 90 days and on a stable dose for 30 days prior to randomization.
* WHO functional class (FC) II or III at randomization
* 6-minute walk distance (6MWD) ≥ 100 m at screening.
* Ability to walk without a walking aid.
* Valid baseline data for daily life physical activity (DLPA) and PAH-SYMPACT®.

Exclusion Criteria:

* Patients on a PAH-specific monotherapy targeting the nitric oxide pathway (i.e. PDE-5 inhibitor or sGC stimulator).
* Patients treated with prostacyclin, prostacyclin analog or selexipag within 3 months prior to screening.
* Any hospitalization during the last 30 days prior to screening.
* Severe coronary heart disease or unstable angina.
* Documented severe hepatic impairment or severe renal insufficiency at screening.
* Participation in a cardio-pulmonary rehabilitation program based on exercise training within 8 weeks prior to screening
* Any factor or condition likely to affect full participation in the study or compliance with the protocol (such as adherence to protocol mandated procedures), as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pfister, Study Director — Actelion
Locations (39):
- United States (15):
  - LA Biomedical Research Institute, Torrance, California
  - Northside Hospital, Atlanta, Georgia
  - Kentuckiana Pulmonary Research Center, Louisville, Kentucky
  - Tufts Medical Center, Pulmonary/Critical Care & Sleep, Boston, Massachusetts
  - University of Nebraska Medical Center, Pulmonary, Critical Care & Sleep Medicine Division, Omaha, Nebraska
  - NYU Winthrop Hospital, Mineola, New York
  - UNC Pulmonary Speciality Clinic, Chapel Hill, North Carolina
  - Duke University School of Medicine, Duke Pulmonary Vascular Disease center, Durham, North Carolina
  - University of Cincinnati, Heart, Lung and Vascular Institute, Cincinnati, Ohio
  - CCF- Akron General Medical Hospital, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Pulmonary Vascular Disease Program, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Care Medicine, Nashville, Tennessee
  - Methodist Clinical Trials, San Antonio, Texas
  - University of Texas Health Science Center (San Antonio), San Antonio, Texas
- Austria (2):
  - Medizinische Universität Innsbruck (MUI), Abt. für Pneumologie, Haus 2, Innsbruck
  - Krankenhaus der Elisabethinen, Servicestelle Klinische Studien, Linz
- France (3):
  - Hôpital Bicêtre, ervice de Pneumologie et Réanimation respiratoire, Le Kremlin-Bicêtre
  - CHRU de Lille - Hôpital Albert Calmette, Service de cardiologie, Lille
  - Hospital Larrey CHU de Toulouse, Toulouse
- Germany (4):
  - Herzzentrum der Universität zu Köln, Klinik III für Innere Medizin, Cologne
  - Universitätsklinikum Giessen, Giessen
  - Universitätsklinikum Leipzig AöR, Abteilung Pneumologie, Leipzig
  - Katholisches Klinikum Lünen/Werne GmbH, Haus E, Lünen
- Mater Misericordiae University Hospital, Dublin, Ireland
- Oslo University Hospital, dept of cardiology, Oslo, Norway
- Portugal (2):
  - Centro Hospitalar e Universitário de Coimbra, Serviço de Cardiologia, Coimbra
  - Hospital Geral de Santo António-DEFI, Porto
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Gothenburg
  - Skåne University Hospital, VO Hjärt och Lungmedicin, Lund
- Switzerland (2):
  - Kantonsspital St. Gallen, Klinik für Pneumologie und Schlafmedizin, Sankt Gallen
  - Universitaetsspital Zurich, Klinik für Pneumologie C HOER 11, Zurich
- United Kingdom (7):
  - Papworth Hospital, Pulmonary Vascular Disease Unit, Cambridge
  - Golden Jubilee National Hospital, Scottish Pulmonary Vascular Unit, Clydebank
  - The Royal Free Hospital, Cardiology Department, London
  - Royal Brompton Hospital, Hypertension, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Cardiothoracic Department, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Pulmonary Vascular Medicine, Sheffield

REFERENCES:
- [Derived] Rehman RZU, Parisi F, Ashraf N, Chatterjee M, Frantz RP, Hemnes AR, Manyakov NV, Carrasco-Zevallos OM, Yardibi T, Selej M, Mansi T, Dunnmon P, Kaliukhovich DA. Characteristics of Daily Walking Bouts as Valid and Reliable Indicators of Exercise Capacity in Pulmonary Arterial Hypertension: Insights From the Randomized Controlled Study With Selexipag (TRACE). Pulm Circ. 2025 May 26;15(2):e70097. doi: 10.1002/pul2.70097. eCollection 2025 Apr. PMID 40433632
- [Derived] Howard LS, Rosenkranz S, Frantz RP, Hemnes AR, Pfister T, Hsu Schmitz SF, Skara H, Humbert M, Preston IR. Assessing Daily Life Physical Activity by Actigraphy in Pulmonary Arterial Hypertension: Insights From the Randomized Controlled Study With Selexipag (TRACE). Chest. 2023 Feb;163(2):407-418. doi: 10.1016/j.chest.2022.08.2231. Epub 2022 Sep 8. PMID 36089068

RESULTS

PARTICIPANT FLOW:
Groups:
- Selexipag: Participants received Selexipag which was up-titrated from Day 1 (Week 1) to Week 12 to the individualized highest tolerated dose (HTD) which ranged from 200 microgram (mcg) to 1600 mcg twice daily (BID) orally. The dose was increased in increments of 200 mcg BID, usually at weekly intervals, depending on the dose tolerability. Up-titration was followed by a stable maintenance treatment period at the highest tolerated dose, from Week 13 to Week 24.
- Placebo: Participants received one to 8 tablets of 200 (mcg) matching placebo, administered up to a maximum dose up-titrated to 1600 mcg orally twice daily. Up-titration was followed by a stable maintenance treatment period at the highest tolerated dose, from Week 13 to Week 24.
Period: Overall Study
Arm/Group | Selexipag | Placebo
Started | 53 | 55
Completed | 50 | 54
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selexipag | Placebo | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14.75) | 49.8 (13.63) | 49.4 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 77
  Male | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 44 | 52 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 0 | 1 | 1
  FRANCE | 2 | 0 | 2
  GERMANY | 6 | 5 | 11
  IRELAND | 1 | 1 | 2
  NORWAY | 0 | 1 | 1
  PORTUGAL | 3 | 3 | 6
  SWEDEN | 4 | 0 | 4
  SWITZERLAND | 0 | 1 | 1
  UNITED KINGDOM | 31 | 35 | 66
  UNITED STATES | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Actigraphy Assessed Daily Life Physical Activity (DLPA) for Variables Expressed in Minutes
Description: Change from baseline to Week 24 of the DLPA activity parameters for daily time spent in non-sedentary activity (NSA) (as defined by Freedson '98 and Koster '16) and daily time spent in moderate-to-vigorous physical activity (MVPA) as defined by Freedson '98 were reported. These variables were assessed by actigraphy and were expressed in minutes. Freedson 1998 established ranges of activity counts obtained from a hip worn accelerometer corresponding to commonly employed MET categories. Based on this work, threshold between sedentary and NSA was defined. This threshold is often referred to as Freedson's 1998 publication. Koster 2016 defined the threshold between sedentary and NSA based on wrist-worn accelerometers on non-dominant hand, respectively. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
minutes
  Daily time spent in NSA (Freedson '98) | -15.2 (79.78) | -25.2 (72.47)
  Daily time spent in MVPA (Freedson '98) | 0.2 (34.48) | -1.9 (34.26)
  Daily time spent in NSA (Koster'16) | -0.7 (72.50) | -15.0 (62.27)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Daily time spent in non-sedentary activity (minutes), Freedson '98; Test type: Other; ANCOVA; Least Square (LS) mean = 13.79, 95% CI 2-sided [13.366 to 40.944], Standard Error of Mean 13.695
Statistical Analysis 2: Comparison: Selexipag vs Placebo; Daily time spent in MVPA (minutes), Freedson '98; Test type: Other; ANCOVA; LS means = 2.31, 95% CI 2-sided [-10.782 to 15.396], Standard Error of Mean 6.601
Statistical Analysis 3: Comparison: Selexipag vs Placebo; Daily time spent in non-sedentary activity (minutes), Koster '16; Test type: Other; ANCOVA; LS mean = 17.81, 95% CI 2-sided [-6.003 to 41.619], Standard Error of Mean 12.008

2. Primary Outcome: Change From Baseline to Week 24 in Actigraphy DLPA for Variables Expressed in Percentage (%)
Description: Change from baseline to Week 24 of the DLPA activity parameters for daily time spent in non-sedentary activity (NSA) (Freedson '98), daily time spent in moderate-to-vigorous physical activity (MVPA) (Freedson '98) and dailytime spent in NSA (Koster '16) were reported. These variables were assessed by actigraphy and were expressed in percentage (%). Freedson 1998 established ranges of activity counts obtained from a hip worn accelerometer corresponding to commonly employed MET categories. Based on this work, threshold between sedentary and NSA was defined. This threshold is often referred to as Freedson's 1998 publication. Koster 2016 defined the threshold between sedentary and NSA based on wrist-worn accelerometers on non-dominant hand, respectively. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: Percentage of daily time spent
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
Percentage of daily time spent
  Daily time spent in NSA (%), Freedson '98 | 0.08 (7.265) | -0.10 (6.439)
  Daily time spent in MVPA (%), Freedson '98 | 0.23 (3.342) | 0.32 (3.513)
  Daily time spent in NSA (%), Koster '16 | 0.80 (7.158) | 0.00 (6.269)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Percentage of daily time spent in non-sedentary activity (%), Freedson '98; Test type: Other; ANCOVA; LS mean = 0.67, 95% CI 2-sided [-1.713 to 3.060], Standard Error of Mean 1.204
Statistical Analysis 2: Comparison: Selexipag vs Placebo; Percentage of daily time spent in MVPA (%), Freedson '98; Test type: Other; ANCOVA; LS mean = -0.05, 95% CI 2-sided [-1.351 to 1.258], Standard Error of Mean 0.658
Statistical Analysis 3: Comparison: Selexipag vs Placebo; Percentage of daily time spent in non-sedentary activity (%), Koster '16; Test type: Other; ANCOVA; LS mean = 1.26, 95% CI 2-sided [-1.104 to 3.618], Standard Error of Mean 1.191

3. Primary Outcome: Change From Baseline to Week 24 in Actigraphy DLPA for Variables Expressed in Counts Per Minute (Counts/Minute)
Description: Change from baseline to Week 24 of the DLPA activity parameter for total daily activities and NSA (Koster '16) were reported. These variables were assessed by actigraphy and were expressed in counts/minutes. Koster 2016 defined the threshold between sedentary and NSA based on wrist-worn accelerometers on non-dominant hand, respectively. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: counts/minute
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
counts/minute
  Total daily activities | 29.3 (337.18) | 18.8 (342.77)
  NSA, Koster '16 | 36.1 (342.11) | 16.8 (351.08)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Volume of total daily activities (counts / minute); Test type: Other; ANCOVA; LS mean = 20.66, 95% CI 2-sided [-105.632 to 146.958], Standard Error of Mean 63.695
Statistical Analysis 2: Comparison: Selexipag vs Placebo; Volume of non-sedentary activity (counts/minute), Koster '16; Test type: Other; ANCOVA; LS means = 27.52, 95% CI 2-sided [-101.945 to 156.976], Standard Error of Mean 65.291

4. Primary Outcome: Change From Baseline to Week 24 in Actigraphy DLPA for Variables Expressed in Counts
Description: Change from baseline to Week 24 of the DLPA activity parameters for volume of non-sedentary activity (Koster '16)were reported. These variables were assessed by actigraphy and were expressed in counts. Koster 2016 defined the threshold between sedentary and NSA based on wrist-worn accelerometers on non-dominant hand, respectively. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
counts | 3898 (345872) | -49187 (343402.2)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Test type: Other; ANCOVA; LS means = 58409, 95% CI 2-sided [-70444 to 187263], Standard Error of Mean 64985

5. Primary Outcome: Change From Baseline to Week 24 in Actigraphy DLPA for Variable Expressed in Step Counts
Description: Change from baseline to Week 24 of the DLPA activity parameters for number of steps during awake time were reported. These variables were assessed by actigraphy and were expressed in step counts. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: step counts
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
step counts | -32.4 (1288.64) | -170.9 (1076.87)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Test type: Other; ANCOVA; LS means = 201.59, 95% CI 2-sided [-242.977 to 646.163], Standard Error of Mean 224.212

6. Primary Outcome: Change From Baseline to Week 24 in Actigraphy DLPA for Variables Expressed in Step Counts/Minute
Description: Change from baseline to Week 24 of the DLPA activity parameters for number of steps during awake time were reported. These variables were assessed by actigraphy and were expressed in step counts/minute. Positive change from baseline means improvement.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The Full Analysis Set (FAS) included all participants randomly assigned to a study treatment.
Measure: Mean (Standard Deviation); unit: step counts/minute
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 53 | 55
step counts/minute | 0.0 (1.25) | 0.0 (1.04)
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Test type: Other; ANCOVA; LS means = 0.07, 95% CI 2-sided [-0.366 to 0.510], Standard Error of Mean 0.221

7. Primary Outcome: Change From Baseline to Week 24 in Total Sleep Time (TST)
Description: TST (in minutes) was assessed by actigraphy.
Time Frame: Baseline and Week 24 (data analysis was done during 14-Days each for Baseline and for Week 24 and mean value reported)
Population: The FAS included all participants randomly assigned to a study treatment. Data was not reported because the sleep episodes were not identified due to unexpected inaccuracy in automated sleep detection algorithm which resulted in missing/unreliable sleep data which would mislead the design of future trials and the interpretation of sleep results.
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change From Baseline to Week 24 in Wake After Sleep Onset (WASO)
Description: WASO (in minutes) was assessed by actigraphy.
Time Frame: Baseline and Week 24 (data collection was done during 14-Days each for Baseline and for Week 24)
Population: as for outcome 7
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Change From Baseline to Week 24 in Number of Awakenings
Description: Number of awakenings was assessed by actigraphy.
Time Frame: Baseline and Week 24 (data collection was done during 14-Days each for Baseline and for Week 24)
Population: as for outcome 7
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change From Baseline to Week 24 in Sleep Efficiency (SE)
Description: SE (in percentage) was assessed by actigraphy. Sleep efficiency was defined as the TST divided by the time in bed (minutes) multiplied by 100. TST was the duration in minutes including REM sleep plus NREM sleep during the time spent in bed.
Time Frame: Baseline and Week 24 (data collection was done during 14-Days each for Baseline and for Week 24)
Population: as for outcome 7
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline to Week 24 in Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Score
Description: PAH-SYMPACT has 2 main parts: symptoms (cardiopulmonary and cardiovascular) and impact (physical impacts and cognitive/emotional). The symptom part is a questionnaire completed daily for 7 consecutive days and contains 11 items. The impact part has a 7-day recall period and is completed on 7th day of symptoms questionnaire data collection period. It contains 11 items pertaining to impact of PAH. The average Cardiopulmonary Symptoms and cardiovascular symptoms domain scores are determined based on daily scores of 6 and 5 items, respectively, reported on a 5-point Likert scale with score range from 0=best to 4=worst. The Physical impacts and Cognitive/emotional domain consists of 7 items reported on a 5-point Likert scale (from 0 to 4). The value 0 = "not at all"/"with no difficulty at all" and value 4 = "very much"/"extremely"/ "not able at all". Mean value on each of 7-day period was calculated for each specific domain score and corresponding mean change from baseline was reported.
Time Frame: Baseline and Week 24
Population: The FAS included all participants randomly assigned to a study treatment. Here, 'N' (Number of participants analyzed) included all participants evaluated for this outcome measure. Here, 'n' (number analyzed) signifies the number of participants evaluable for a specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 44 | 52
units on a scale
  Cardiopulmonary symptoms | -0.030 (0.4160) | -0.080 (0.2564)
  Cardiovascular symptoms | 0.010 (0.3522) | -0.045 (0.3029)
  Physical impact: number analyzed (Participants) | 40 | 50
  Physical impact | -0.043 (0.5932) | -0.074 (0.5470)
  Cognitive/emotional impact: number analyzed (Participants) | 40 | 50
  Cognitive/emotional impact | 0.000 (0.5311) | -0.090 (0.5992)

12. Secondary Outcome: Number of Participants With Change From Baseline to Week 24 in World Health Organization Functional Class (WHO FC)
Description: The WHO FC of pulmonary hypertension is a physical activity rating scale as follows: Class I (No limitation of physical activity); Class II (Slight limitation of physical activity); Class III (Marked limitation of physical activity); and Class IV (Inability to carry out any physical activity without symptoms). The change from baseline in WHO FC was classified into "Improved", "No change" and "Worsened" compared to baseline. Deterioration, No Change, and Improvement are based on shift of risk category (I, II, III, IV) from baseline in WHO Functional Class.
Time Frame: Baseline and Week 24
Population: The FAS included all participants randomly assigned to a study treatment. Here 'N' (number of participants analyzed) included all participants who were with assessments at both baseline and post-baseline time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 44 | 52
Participants
  Deterioration | 2 | 1
  No change | 33 | 43
  Improvement | 9 | 10

13. Secondary Outcome: Change From Baseline to Week 24 in 6-Minute Walk Distance (6MWD)
Description: The 6MWD was the total distance walked during 6 minutes. Mean change from baseline (distance walked at Week 24 minus distance walked at baseline) was reported.
Time Frame: Baseline and Week 24
Population: The FAS included all participants randomly assigned to a study treatment. Here, N (Number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 50 | 54
meters | 18.3 (54.47) | 9.8 (60.72)

14. Secondary Outcome: Change From Baseline to Week 24 in Borg Dyspnea Score
Description: The Borg dyspneas score was a self-rating scale to evaluate the severity of dyspnea (from 0 "no shortness of breath at all" to 10 "very, very severe / maximal") shortness of breath. It was completed immediately after the 6-minute walk test at Week 24 and at baseline. Mean change from baseline in scoring was reported.
Time Frame: Baseline and Week 24
Population: The FAS included all participants randomly assigned to a study treatment. Here, N (Number of Participants Analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 50 | 54
units on a scale | -0.25 (2.122) | 0.37 (1.869)

15. Secondary Outcome: Change From Baseline to Week 24 in N-Terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: Change from baseline to Week 24 in NT-pro BNP levels was reported. The negative change from baseline means improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 51 | 53
nanogram per liter (ng/L) | -153.8 (609.32) | 81.8 (316.54)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: Safety Analysis Set included the participants who were who were randomized and received at least 1 dose of study treatment.
Arm/Group | Selexipag | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/53 | 6/55
Other Adverse Events (participants affected / at risk) | 52/53 | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=53) | Placebo (N=55)
Atrial Flutter (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Vision Blurred (Eye disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thyroid Nodule Removal (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=53) | Placebo (N=55)
Palpitations (Cardiac disorders) | 2 | 4
Abdominal Distension (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 28 | 23
Dyspepsia (Gastrointestinal disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 22 | 15
Vomiting (Gastrointestinal disorders) | 13 | 4
Fatigue (General disorders) | 5 | 4
Non-Cardiac Chest Pain (General disorders) | 2 | 7
Oedema Peripheral (General disorders) | 3 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 14
Respiratory Tract Infection (Infections and infestations) | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 6
Urinary Tract Infection (Infections and infestations) | 0 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 20 | 5
Dizziness (Nervous system disorders) | 7 | 7
Headache (Nervous system disorders) | 41 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Flushing (Vascular disorders) | 5 | 6
Hot Flush (Vascular disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
No hypothesis testing was planned for this exploratory study. Data for sleep outcome measures were not reported because the sleep episodes were not identified due to unexpected inaccuracy in automated sleep detection algorithm which resulted in missing/unreliable sleep data which would mislead the design of future trials and the interpretation of sleep results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, Actelion may provide comments and may also request alterations and/or deletions for the sole purpose of protecting its confidential information or patent rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03078907/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03078907/SAP_001.pdf